CLINICAL TRIAL: NCT05971342
Title: A Two-arm Clinical Study to Evaluate the Safety and Efficacy of Gelatin Sponge-loaded Apoptotic Vesicle Complex for Alveolar Bone Defect Repair After Mandibular Third Molar Extraction
Brief Title: The Safety and Efficacy of Alveolar Bone Defect Repair Induced by Gelatin Sponge-loaded Apoptotic Vesicle Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mao Xue Li
Record Dates: First submitted 2023-06-14; First posted 2023-08-02 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2023-07

CONDITIONS: Third Molar Extraction
Keywords: Third Molar Extraction; Alveolar Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gelatin sponge-loaded apoptotic vesicle complex (Experimental): 4 * 10^10 apoptotic vesicles derived from umbilical cord mesenchymal stem cells were loaded in a gelatin sponge（Kuaikang®）. A piece of gelatin sponge-loaded apoptotic vesicle complex was placed in an extraction socket after tooth extraction.
  Interventions: Drug: Gelatin sponge-loaded apoptotic vesicle complex（Kuaikang®)
- Gelatin sponge only (Active Comparator): A piece of gelatin sponge（Kuaikang®）was placed in an extraction socket after tooth extraction.
  Interventions: Drug: Gelatin sponge only （Kuaikang®)

INTERVENTIONS:
Drug: Gelatin sponge-loaded apoptotic vesicle complex（Kuaikang®) — The experimental group
  Other Names: Gelatin sponge （Kuaikang®）. Apoptotic vesicles are derived from umbilical cord mesenchymal stem cells
  Arms: Gelatin sponge-loaded apoptotic vesicle complex
Drug: Gelatin sponge only （Kuaikang®) — The positive control group
  Other Names: Gelatin sponge （Kuaikang®）
  Arms: Gelatin sponge only

SUMMARY:
Distal bone loss of the second molar due to extraction of the third molar is one of the most common pathological conditions that results in tooth loss of second molar. However, regeneration of functional alveolar bone has proved difficult. Therefore, the investigators conduct a two-arm study to evaluate the efficacy and safety of alveolar bone regeneration induced by gelatin sponge-loaded apoptotic vesicle complex in patients with mandibular third molar extraction.

DETAILED DESCRIPTION:
This study is a single-center, prospective, two-arm study to evaluate the efficacy and safety of alveolar bone regeneration induced by gelatin sponge-loaded apoptotic vesicle complex in patients with mandibular third molar extraction. This study plans to include 30 subjects from the Department of Stomatology of the Fifth Affiliated Hospital of Guangzhou Medical University. One socket for each participant in this study will receive gelatin sponge-loaded apoptotic vesicle complex after third molar extraction and socket debridement. The other side of socket for each participant in this study will receive commercial gelatin sponge after the same surgery. All participants will undergo screening and baseline visits. After surgery, the participants will be followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-45 (including the boundary value)
2. Patients who need to extract the bilateral mandible third molars
3. Patients who voluntarily sign the informed consent form

Exclusion Criteria:

1. The adjacent second molars in the patient's oral cavity are affected by pulp injury or insufficient endodontic treatment, or show tooth fracture, or have a degree of motion of 3 degrees
2. The adjacent second molars have metal crowns or large amalgam restorations
3. There is an uncontrollable pathological process in the patient's oral cavity
4. Malnutrition (serum albumin concentration <2 g/dl)
5. Other systemic, infectious diseases and hereditary diseases, or patients in the acute inflammatory phase and acute exacerbation phase of chronic diseases
6. Patients who are pregnant, lactating, or planning to become pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Bone volume fraction of regenerated bone tissue in the extraction area at 3 months after operation | 3 months
  CBCT is a cone-beam projection computerized reconstruction tomography device. Its principle is that the X-ray generator uses a low radiation dose to make a circular DR (digital projection) around the projection body. Then the data obtained in the "intersection" after digital projection around the projection body multiple times is "reconstructed" in the computer to obtain a three-dimensional image. CBCT can observe the three-dimensional level of bone regeneration, so as to calculate the bone volume fraction of the regenerated bone tissue.

SECONDARY OUTCOMES:
Hemostatic time after third molar extraction | 0 day
  After the third molar was completely extracted, commercial gelatin sponge or gelatin sponge loaded with apoptotic vesicle complex were placed in the socket. The time to hemostasis in the extraction socket was observed and recorded at the same time.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No